CLINICAL TRIAL: NCT05076734
Title: Technology Development for Noninvasive Prenatal Genetic Diagnosis Using Maternal Peripheral Blood: N o Return of Results -Luna Collection
Brief Title: Cell- Based Noninvasive Prenatal Testing (NIPT): Single Cell Prenatal Diagnosis (SCPD)
Acronym: NIPT & SCPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luna Genetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Luna IRB LG-002
Record Dates: First submitted 2021-09-16; First posted 2021-10-13 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Analysis of blood samples from healthy pregnant women (Other): A phlebotomist will be sent to any location in the United States to collect the blood sample. Sample identifiers will be removed as the first step so that laboratory personnel will not see or have access to identifiers. No information will go back to patients or their physicians.
  Interventions: Diagnostic Test: Redraw for analysis of blood samples from healthy pregnant women

INTERVENTIONS:
Diagnostic Test: Redraw for analysis of blood samples from healthy pregnant women — If less than two fetal cells are recovered from maternal blood, a redraw is indicated

SUMMARY:
The purpose of the overall study is to develop improved methods for recovery of fetal cells from the mother's blood in order to develop a clinically useful form of cell-based, diagnostic, noninvasive prenatal testing (NIPT). Luna Genetics will analyze blood samples from healthy pregnant women. A phlebotomist will be sent to any location in the United States to collect the blood sample. Sample identifiers will be removed as the first step so that laboratory personnel will not see or have access to identifiers. No information will go back to patients or their physicians.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* 18years or older

Exclusion Criteria:

* Language barrier (non-English speaking and no adequate interpreter)
* Maternal age of less than 18 years
* Higher order multiple pregnancy (triplet or greater)
* Not currently pregnant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females, 18 years and older
Enrollment: 157 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Fetal Cell Recovery and genetic analysis | 2 months
  Outcome 1 is the number of cells identified as fetal by microscopic staining. This can be converted to units based on volume. If 40 mL of blood is collected and f8 cells are designated as fetal based on microscopic staining, the results can be tabulated as follow: So a result is 8 cells are identified as fetal from one blood draw. This equals 0.2 cells identified per mL of maternal blood. If two or fewer cells are obtained, a blood redraw will be requested from the patient.
Redraw for Fetal Cell Recovery and genetic analysis | 2 months
  Outcome measure 2 is the number of cells that yield high quality next generation sequencing data suitable for determining copy number across the entire genome. So if 4 of the 8 cells above gave high quality data, the outcome would be 4 cells with high quality copy number data from one blood draw which equals 0.10 high quality cell / mL of mother's blood.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Beaudet, MD, Principal Investigator — Luna Genetics
Locations (1):
- Luna Genetics, Houston, Texas, United States